CLINICAL TRIAL: NCT05844059
Title: Lower Urinary Tract Symptoms After Intravesical Therapy With Mitomycin C or BCG in Patients With Carcinoma of the Bladder
Brief Title: Lower Urinary Tract Symptoms After Intravesical Therapy
Acronym: LUTSI
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Benedikt Ebner, Dr. med., Ludwig-Maximilians - University of Munich
Other Study IDs: 23-0226
Record Dates: First submitted 2023-04-22; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chemotherapy Effect; Chemotherapeutic Toxicity; Lower Urinary Tract Symptoms; Overactive Bladder
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing instillation therapy with BCG: All patients that undergo therapy with BCG after diagnosis of non-muscle-invasive bladder cancer
  Interventions: Other: Validated questionnaires
- Patients undergoing instillation therapy with Mitomycin C: All patients that undergo therapy with Mitomycin C after diagnosis of non-muscle-invasive bladder cancer
  Interventions: Other: Validated questionnaires

INTERVENTIONS:
Other: Validated questionnaires — BPIC-SS, ICIQ-OABqol, IIEF-EF oder FSFI, ICIQ-MLUTS oder ICIQ-FLUTS

SUMMARY:
With this prospective, observational study, we would like to investigate the effect of instillation therapy using BCG or mitomycin C on short- and long-term irritative and obstructive lower urinary tract symptoms using validated questionnaires. The study will objectify the lower urinary tract symptoms and thereby provide better recommendations for therapy with mitomycin C or BCG.

ELIGIBILITY:
Inclusion Criteria:

* Urinary bladder carcinoma requiring instillation therapy
* Complete resection of the tumor
* No intravesical chemotherapy in the last 3 months

Exclusion Criteria:

* Patients who are unable to complete the questionnaires
* Patients who are not willing to participate
* Patients with contraindications for instillation therapy (allergic reactions, immunosuppression)

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with urinary bladder carcinoma requiring instillation therapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Effect of instillation therapy on quality of life | During the study period approximately 12 months
  Quality of life will be measured with validated questionnaires such as the ICIQ-OABqol
Effect of instillation therapy on sexuality | During the study period approximately 12 months
  Sexuality will be measured with validated questionnaires such as the IIEF-EF (men) and the FSFI (women)
Effect of instillation therapy on lower urinary tract symptoms | During the study period approximately 12 months
  Lower urinary tract symptoms will be measured with validated questionnaires such as the BPIC-SS, the ICIQ-MLUTS (men) and the ICIQ-FLUTS (women)

SECONDARY OUTCOMES:
Complications during instillation therapy | During the study period approximately 12 months
  The frequency of all complications will be measured and will be subsequently classified based on the Clavien-Dindo classification
Discontinuation rate of instillation therapy | During the study period approximately 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nikolaos Pyrgidis, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No